CLINICAL TRIAL: NCT01213732
Title: Phase 1 Dose-finding Study of Tumor-targeting Human Monoclonal Antibody-cytokine Fusion Protein L19TNFα Plus Melphalan Using Isolated Inferior Limb Perfusion in Patients With In-transit Stage III/IV Melanoma.
Brief Title: Phase 1 Dose-finding Study of L19TNFα Plus Melphalan Using Isolated Inferior Limb Perfusion (ILP) in Subjects With Intransit Stage III/IV Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Philogen S.p.A. (Industry)
Collaborators: InnoPharma Inc. (Industry); Eudax S.r.l. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PH-L19TNFαILP-01-08
Record Dates: First submitted 2010-10-01; First posted 2010-10-04 (Estimated); Last update posted 2022-04-15 (Actual); Status verified 2011-09

CONDITIONS: Patients With Intransit Stage III/IV Melanoma
Keywords: L19, antibody, monoclonal, tumor targeting, TNFa, ILP, melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- L19TNFα plus melphalan (Experimental): Subjects will be sequentially assigned to one of 2 dose levels of L19TNFα: 325 µg or 650 µg. All subjects will receive a single dose of L19TNFα and Melfalan (10mg/ L Limb volume).
  Interventions: Other: Isolated inferior limb perfusion

INTERVENTIONS:
Other: Isolated inferior limb perfusion — Single Melphalan bolus perfused for 60 min after 30 min of L19TNFα bolus. Intra-arterial (IA) infusion via bolus at 39˚C to 40˚C (mild hyperthermia).

SUMMARY:
In this study the recombinant human fusion protein L19TNFα will be associated in ILP with the standard treatment with melphalan 10mg/l limb volume in subjects affected by stage III/IV limb melanoma.

The recombinant human fusion protein L19TNFα was created with the intention to target TNFα directly to tumor tissues with the result in high and sustained intralesional bioactive TNFα concentrations.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged >18 years.
2. Histologically or cytologically confirmed intransit stage III/IV melanoma of lower extremity distal to the apex of the femoral triangle
3. ECOG performance status ≤ 2.
4. Subjects must have at least one unidimensional clinically measurable lesion as defined by RECIST criteria (see Section 8). This lesion must not have been irradiated within four weeks during previous treatments.
5. Absolute neutrophil count (ANC) ≥ 1.5 x 109/L, platelets ≥ 100 x 109/L, and haemoglobin (Hb) ≥ 9.5 g/dl.
6. All acute adverse effects (excluding alopecia) of any prior therapy (including surgery, radiation therapy, chemotherapy) must have been resolved to ≤ Grade 1, except elevated liver transaminases judged to be associated with tumor infiltration (see below) (graded according to National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events, version 3.0 [CTCAE, v.3.0].
7. Alkaline phosphatase (AP), alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) ≤ 2.5 x upper limit of normal (ULN), and total bilirubin ≤ 2.0 mg/dL unless liver involvement by the tumor, in which case the transaminase levels up to 5 x ULN are allowed.
8. Creatinine ≤ 1.5 ULN or 24 h creatinine clearance ≥ 60 mL/min.
9. Testing negative for acute or chronic infection with hepatitis B or C virus, or human immunodeficiency virus 1 or 2.
10. Negative pregnancy test for females of childbearing potential at the screening visit.
11. Commitment from subject to practice medically appropriate/acceptable method of birth control (e.g., hormonal, condoms or other adequate barrier controls, intrauterine contraceptive device, or sterilization) beginning at the screening visit and continuing until 3 months following the treatment with study drug
12. Able to provide written Informed Consent
13. Willingness and ability to comply with the scheduled visits, treatment plan, laboratory tests and other study procedures.

Exclusion Criteria:

1. Breastfeeding women
2. Presence of active infections (e.g. requiring antimicrobial therapy) or other severe concurrent disease, which, in the opinion of the Investigator, would place the subject at undue risk or interfere with the study.
3. Active autoimmune disease.
4. Cardiac disease as manifested by any of the following:

   * > Grade II heart failure, graded per New York Heart Association (NYHA) criteria.
   * Unstable angina pectoris
   * Acute or subacute coronary syndromes, including myocardial infarction, occurring with 1 year prior to study treatment
   * Arrhythmia needing continuous treatment
   * Ejection fraction less than the institutional lower limit of normal as assessed by multigated radionuclide angiography (MUGA) scan or echocardiogram
5. Uncontrolled hypertension.
6. History of claudication or Ischemic peripheral vascular disease (Grade IIb-IV).
7. Chronic obstructive pulmonary disease or other chronic pulmonary disease with PFTs less than 50% predicted for age.
8. Symptomatic cerebrovascular disease.
9. Active peptic ulcer disease.
10. Concurrent infection of HIV.
11. Severe diabetic retinopathy.
12. Major surgery or trauma within 4 weeks prior to start of study treatment.
13. Hypersensitivity to melphalan or TNFα or other intravenously administered human proteins/peptides/antibodies.
14. Chemotherapy, radiation therapy or therapy with an investigational agent within 4 weeks prior to start of study treatment.
15. Any regional therapy to the affected extremity within 2 months prior to start of study treatment.
16. Previous in vivo exposure to monoclonal antibodies for biological therapy in the 6 weeks before administration of study treatment.
17. Growth factors or immunomodulatory agents within 7 days prior to the administration of study treatment.
18. Subject requires or is taking corticosteroids or other immunosuppressant drugs on a long-term basis. Limited use of corticosteroids to treat or prevent acute hypersensitivity reactions is not considered an exclusion criterion.
19. Participation in another interventional clinical trial during participation in this trial.
20. Any conditions that in the opinion of the Investigator could hamper compliance with the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2008-10; Primary Completion 2011-03 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability | 6 weeks
  The safety and tolerability profile of L19TNFα/melphalan combination treatment in the ILP setting will be determined.
Recommended dose (RD) | 29 days
  The recommended dose (RD) of L19TNFα when given in combination with melphalan in the ILP setting for subjects with limb stage III/IV melanoma will be determined.

SECONDARY OUTCOMES:
Objective response rate | 10 weeks
  Objective response rate of L19TNFα plus melphalan.
Antitumor activity | 4- 6 weeks
  Antitumor activity of L19TNFα plus melphalan (resection of residual tumor after 4- 6 weeks and histopathological response rate).
Pharmacokinetic | 10 days
  Pharmacokinetic profile of L19TNFα when given with melphalan
Human anti-fusion protein antibody | 6 weeks
  Assessment of possible induction of human anti-fusion protein antibody [HAFA] formation
5-hydroxyindoleacetic acid | 10 days
  Assessment of plasma profile of 5-hydroxyindoleacetic acid (5-HIAA), a surrogate marker of vascular damage and tumor response.

CONTACTS AND LOCATIONS:
Overall Officials: Franco De Cian, Prof, Principal Investigator — IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy
Locations (2):
- Italy (2):
  - Azienda Ospedaliera Universitaria San Martino, Genova
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan

REFERENCES:
- [Derived] Papadia F, Basso V, Patuzzo R, Maurichi A, Di Florio A, Zardi L, Ventura E, Gonzalez-Iglesias R, Lovato V, Giovannoni L, Tasciotti A, Neri D, Santinami M, Menssen HD, De Cian F. Isolated limb perfusion with the tumor-targeting human monoclonal antibody-cytokine fusion protein L19-TNF plus melphalan and mild hyperthermia in patients with locally advanced extremity melanoma. J Surg Oncol. 2013 Feb;107(2):173-9. doi: 10.1002/jso.23168. Epub 2012 Jun 4. PMID 22674435